CLINICAL TRIAL: NCT05120882
Title: Epidemiology of Lupus Nephritis in Nephrology Unit in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ekram Farouk Ibrahim, Lupus nephritis patients in Nephrology Unit in assiut University hospital, Assiut University
Other Study IDs: lupus nephritis
Record Dates: First submitted 2021-10-30; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
study epidemiology of lupus nephritis patients admitted to nephrology unit inward or in outpatient clinic in Assiut Nephrology Unit

DETAILED DESCRIPTION:
this study are:

To describe socio-demographic characteristics of lupus nephritis patients in Nephrology Unit of Assiut University hospital ( Old and New cases).

To determine the associated risk factors in the study population

To describe the clinical, laboratory characteristics, treatment modalities of lupus nephritis patients in Nephrology Unit of Assiut University hospital ( Old and New cases)

To Identify outcomes of treatment of these cases within 2 years according to different classes

To evaluate the effectiveness of (type of interventions mentioned) among those patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to nephrology unit or visiting the outpatient nephrology clinic,previously or newly diagnosed with lupus nephritis.

Exclusion Criteria:

* incomplete Criteria for diagnosis of systemic lupus or presence of associated renal disease.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to nephrology unit or visiting the outpatient nephrology clinic, previously or newly diagnosed with lupus nephritis in Internal Medicine Department in assiut University hospital will be recruited from December 2021 till May 2022.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Study of epidemiology of lupus nephritis patients | 6 months
  Detection of different risk factors such as socioeconomic status and its relation to lupus nephritis To study the outcome of treatment plans in different classes of lupus nephritis